CLINICAL TRIAL: NCT03021005
Title: Provision of HIV Self-Test Kit to Increase Uptake of HIV Testing Among Emergency Department Patients Who Decline Emergency Department-Based HIV Screening.
Brief Title: Provision of HIV Self-Test Kit to Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00090921; U54EB007958 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self Testing Kit (Experimental): This group will be provided a free Food and Drug Administration-approved HIV self-testing home kit (OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test). Participants in this group will also be provided 5 referral cards to give to their partners and peers in the drug, sex, and social networks for them to request a free HIV self-testing kit from the "I Want The Kit" website.
  Interventions: Behavioral: HIV Self-testing
- No Self Testing Kit (No Intervention): This group will not receive a free Food and Drug Administration-approved HIV self-testing home kit (OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test). Participants in this group will not receive referral cards for their partners or peers for them to request a free HIV self-testing kit from the "I Want The Kit" website.

INTERVENTIONS:
Behavioral: HIV Self-testing
  Arms: Self Testing Kit

SUMMARY:
The proposed pilot research has three aims: 1) to determine the feasibility and acceptability of provision of HIV self-testing kit in order to increase uptake and engagement of HIV testing among emergency department patients who decline conventional emergency department HIV testing and to increase the engagement of HIV testing at a regular basis for those with an increased risk for HIV (the index participants); 2) to determine the uptake and engagement of HIV testing by provision of HIV self-testing kit; and 3) to determine the feasibility and acceptability of HIV self-testing kit referral among partners or peers of the index participants.

The investigators will conduct a pilot randomized study at Johns Hopkins Hospital emergency department on (1) patients who decline routine HIV testing offer and (2) patients who are at an increased risk for HIV. The consented patient will be randomized to HIV self-testing kit group which the investigators will provide a free Food and Drug Administration-approved HIV self-testing home kit for the participant to take it home or to reference group which the investigators will not provide the self-testing kit. Consented patients in both groups will fill out a short survey regarding their socio-demographic information as well as their experience and perceptions regarding HIV testing. For patients who are in the HIV self-testing kit group, they will be asked if they would like to take a free HIV self-testing home kit home. Participants in this group will also receive information regarding how to access "I Want The Kit" website to report the completion of HIV self-testing at home. For patients who are in the reference group, a standard pamphlet regarding the importance of HIV testing and HIV testing venues in Baltimore City used by emergency department-based HIV testing program will be provided to the patients.

Follow-up questionnaires will inquire regarding the patient's experience regarding HIV testing since their index visit.

When the participants in the HIV self-testing kit group in Aim 1, they will also be provided 5 referral cards for their partners and peers for them to request a free HIV self-testing kit from the "I Want The Kit" website. At the 1-month phone follow-up, the investigators will ask participants if they are able to give the referral cards to their partner(s) or friend(s), how they think if their partner(s) and/or friend(s) will request an HIV self-testing kit from the "I Want The Kit" website.

DETAILED DESCRIPTION:
The Investigators will conduct a pilot randomized study at Johns Hopkins Hospital Emergency Department on patients who decline routine HIV testing offer by triage nurses. 1. Recruitment

"Refusers" Cohort Study staff will screen the emergency department tracking board (Epic) for patients who meet study enrollment criteria, which is done routinely as part of the emergency department HIV testing program. When an eligible patient is identified by the chart review (please see HIPAA form 4), the study staff will talk to the emergency department clinician regarding research opportunity for the potentially eligible patients. For all individuals who are not clinical patients of a study team member, the recruitment procedure will be that the patient's clinician will request and document in the chart the patient's permission to be contacted by the research staff.

"High Risk" Cohort "The eligibility of "high-risk cohort" is emergency department patients who are offered an HIV test as the standard of care in the emergency department, accept the standard of care (SOC) HIV testing, and who have at increased risk for HIV. Study staff will screen the emergency department tracking board (Epic) for patients who are offered an HIV test at triage by the triage nurse, which is done routinely as part of the emergency department HIV testing program. When an eligible patient is identified by the chart review (please see HIPAA form 4), the study staff will talk to the emergency department clinician regarding research opportunity for the potentially eligible patients. For all individuals who are not clinical patients of a study team member, the recruitment procedure will be that the patient's clinician will request and document in the chart the patient's permission to be contacted by the research staff. In order to determine if the patient is at increased risk for HIV, the study staff will use of the Screening Question (three screening questions) that is uploaded in the application section 20 (see section 20 for Screening_Question_05312016"). The three questions are as follows: 1) Have you been sexually active in the past 12 months, 2) have you ever used injection drugs in your life, and 3) (for men only), have you ever had sex with a man in your life time. If the patient responds "yes" to the question "Is any of your answer "Yes" (see section 20 for Screening_Question_05312016"), they will be considered eligible and will then go through the consent and enrollment procedures. No identifiers will be collected for this screening step.

2. Enrollment The study staff will obtain verbal informed consent. The process will involve a description of the study as provided in the verbal consent form (OralConsentScript_for_HighRiskPatient_06012016.docx) with a chance to provide answers to any questions about the study. Justification for verbal consent is provided in the e-Institutional Review Board application. Specifically, this study involves no bodily intervention and poses minimal risk to patients. The consent process will take between approximately 5-10 minutes, but as much time as needed will be provided to patients. Consented subjects will be given a copy of the oral

consent document for their information and records. In this consent, the patient will be asked for permission to review their medical charts at Johns Hopkins Hospital for the clinical information of their emergency department visit. Consented patients will be randomized to one of two groups, the Index Group (Group 1) or the Reference Group (Group 2). The index group or the HIV self-testing kit group will be provided a free FDA-approved HIV self-testing home kit (OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test) and the reference group will not receive the HIV self-testing kit. Consented patients in both groups will fill out a short survey regarding their socio-demographic information as well as their experience, attitudes, and perceptions regarding HIV testing. For patients who are in the HIV self-testing kit group, they will be asked if they would like to take a free FDA-approved HIV self-testing home kit home. If they agree, the research staff will make sure the patients will take the kit home when they are discharged. Participants in this group will also receive information regarding how to access the "I Want The Kit" website to report the completion of HIV self-testing at home. Participants in this group will also be informed of a lottery-based monetary compensation with 1 in 10 chance to win an additional $50 gift card for reporting the test results to the "I Want The Kit" website. Participant who wins the $50 gift card will be notified via text message, followed by a phone call while participant who does not win the gift card will be notified via text message (see section 20 for "Text Message Script for Lottery Incentive). For patients who are in the reference group, a standard pamphlet regarding the importance of HIV testing and HIV testing venues in Baltimore City used by current Johns Hopkins Hospital emergency department-based HIV testing program will be provided to the patients.

3. Survey information:

* Patients will be consented and enrolled in the study prior to collecting data in the emergency department.
* After patient consent and enrollment by the study staff, each study participant will complete a survey questionnaire (see attached Index_Questionnaire.docx in Supplemental Study Documents) at the time of enrollment to indicate their social, demographic, and clinical characteristics. The survey is research (not part of routine care), but would not add to the patient's length of stay since it can be conducted during waiting time in a private setting. This survey will be clearly explained by and completed with the assistance of the study staff.
* All patients will be informed of intent to contact them for a brief follow-up phone interview at one month and 3 months from the date of enrollment. This is one of the exclusion criteria.
* Following enrollment, a member of the research team will abstract chart data of the emergency department visits. The abstraction will focus on visit-specific clinical data (e.g. chief complaint, diagnosis, acuity level, and disposition (The full variable list can be found in section 20, Variable List).

  4. Patient Follow-up
* Participants will receive a phone or text message reminder from the study team in order to remind that they are enrolled in the study within a week after the enrollment. The study team will make sure that the participant is the one who answers the phone before reminding the participant of this study. The text message will not contain the words of HIV or HIV testing. The participant will also receive text message reminder 1 week before each follow-up time (1 and 3 month time point). The text message will include the reminder of the phone follow-up as well as the $10 gift card incentive that the investigators would be providing to the participant upon completing the phone follow up (see section 20 for "Text reminder version 0.02).
* Consented patients will be contacted by the study team at one month and 3 months after enrollment. No more than five separate attempts to contact will be made during this time until deemed lost to follow up for the particular follow up time point.
* Follow-up questionnaires will ask the patient about their experience, attitudes, and perceptions regarding HIV testing since their index visit. Please see attached Phone_Script.docx
* A $10.00 gift card will be mailed to the participant once he/she completes the follow-up survey by phone for each follow up time point.

  5. HIV Self-testing at home Instructions for performing the home test, with visual aids, will be included with the kit. For participants in the HIV self-testing kit group whose test result by HIV self-testing at home is interpreted as "reactive" or "indeterminate", he or she can follow the instruction inside the kit to call a hotline to Johns Hopkins Hospital emergency department routine rapid HIV screening and linkage to care program staff that operates 16 hours a day, 7 days a week, OraQuick Consumer Support Center that operates 24 hours a day, or their primary physician for counseling. Patients with a reactive test result can either come to Johns Hopkins Hospital emergency department or the Johns Hopkins HIV Women's Program to receive confirmatory blood testing of the screening self-test. All participants with a positive or indeterminate screening result will have blood drawn and sent to the Maryland Department of Health and Mental Hygiene Laboratories Administration Central Laboratory where free confirmatory testing will be performed using the HIV-1 Western Blot Assay from Bio-Rad Laboratories. (At Maryland Department of Health and Mental Hygiene and Central Laboratory, indeterminate and negative HIV-1 Western Blot specimens are tested using the Multispot HIV-1/HIV-2 Rapid test as a differentiation assay to rule out HIV-2, and using in-house validated HIV-1 real time polymerase chain reaction assay to detect acute cases of HIV-1).

For participants in the HIV self-testing kit group, they will be asked to report their test result on to "I Want The Kit" website using the access information provided in the HIV self-testing kit.

When the participants (the index participants) in the HIV self-testing kit group in Aim 1 receive the self-testing kit, they will also be provided 5 referral cards to give to their partners and peers in the drug, sex, and social networks for them to request a free HIV self-testing kit from the "I Want The Kit" website. On the referral card, a unique code number be used after the subject uses provided website address to land in "I Want The Kit" website and create an "I Want The Kit" user account. The unique code number will indicate the "I Want The Kit" user is referred from an emergency department patient who is an index participant. The index participants would also be informed of a lottery-based monetary compensation to provide 1 in 10 chance to win an additional $10 gift card for every "I Want The Kit" user that is referred from an index participant of this study. Participant who wins the $10 gift card will be notified via text message, followed by a phone call while participant who does not win the gift card will be notified via text message (see section 20 for "Text Message Script for Lottery Incentive). The confidential code numbers will allow determination of whether emergency department subjects and/or their referrals use the "I Want The Kit" website but will not allow research team access to identity-linked test results (Please see data management section below regarding de-identification before data analysis). At the 1-month and 3-month phone follow-up, the investigators will ask participants if they are able to give the referral cards to their partner(s) or friend(s), how many cards they are able to give out, how many cards they are able to give to their partner(s), how many cards they are able to give to their friend(s), and how likely it is that their partner(s) and/or friend(s) will request an HIV self-testing kit from the "I Want The Kit" website. Finally, the investigators will ask them how the investigators can increase the likelihood of their partner(s) and/or friend(s) accessing the "I Want The Kit" website and requesting an HIV self-testing kit.

ELIGIBILITY:
Inclusion Criteria:

* Johns Hopkins Hospital emergency department patients who decline routine HIV testing offer ("Decliners") or patients who are offered an HIV test as the standard of care in the emergency department , accept the standard of care (SOC) HIV testing, and who have at increased risk for HIV "High Risk").

Exclusion Criteria:

* Any person who is already known to be HIV positive. Patients with a chief complaint of sexual assault, patients with chief complaint of occupational exposure and patients who are otherwise ineligible to consent to an HIV test due to medical condition (e.g., severe illness, altered mental status). Any person who has previously enrolled in this study. Any person less than 18 years of age. Any person who is not able to provide contact information for follow-up survey. Any person who reports they are unable to access the internet.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Hsieh, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Branson BM, Handsfield HH, Lampe MA, Janssen RS, Taylor AW, Lyss SB, Clark JE; Centers for Disease Control and Prevention (CDC). Revised recommendations for HIV testing of adults, adolescents, and pregnant women in health-care settings. MMWR Recomm Rep. 2006 Sep 22;55(RR-14):1-17; quiz CE1-4. PMID 16988643
- [Background] Centers for Disease Control and Prevention (CDC). Missed opportunities for earlier diagnosis of HIV infection--South Carolina, 1997-2005. MMWR Morb Mortal Wkly Rep. 2006 Dec 1;55(47):1269-72. PMID 17136020
- [Background] Czarnogorski M, Brown J, Lee V, Oben J, Kuo I, Stern R, Simon G. The Prevalence of Undiagnosed HIV Infection in Those Who Decline HIV Screening in an Urban Emergency Department. AIDS Res Treat. 2011;2011:879065. doi: 10.1155/2011/879065. Epub 2011 May 9. PMID 21738860
- [Background] Johnson C, Baggaley R, Forsythe S, van Rooyen H, Ford N, Napierala Mavedzenge S, Corbett E, Natarajan P, Taegtmeyer M. Realizing the potential for HIV self-testing. AIDS Behav. 2014 Jul;18 Suppl 4:S391-5. doi: 10.1007/s10461-014-0832-x. PMID 24986599
- [Background] Vargo S, Agronick G, O'Donnell L, Stueve A. Using peer recruitment and OraSure to increase HIV testing. Am J Public Health. 2004 Jan;94(1):29-31. doi: 10.2105/ajph.94.1.29. PMID 14713690
- [Background] Gaydos CA, Hsieh YH, Harvey L, Burah A, Won H, Jett-Goheen M, Barnes M, Agreda P, Arora N, Rothman RE. Will patients "opt in" to perform their own rapid HIV test in the emergency department? Ann Emerg Med. 2011 Jul;58(1 Suppl 1):S74-8. doi: 10.1016/j.annemergmed.2011.03.029. PMID 21684413
- [Background] Nour S, Hsieh YH, Rothman RE, Jett-Goheen M, Langhorne O, Wu L, Peterson S, Gaydos CA. Patients Can Accurately Perform Their Own Rapid HIV Point-of-Care Test in the Emergency Department. Point Care. 2012 Dec 1;11(4):176-179. doi: 10.1097/POC.0b013e3182666eb7. PMID 24031999
- [Background] Chai SJ, Aumakhan B, Barnes M, Jett-Goheen M, Quinn N, Agreda P, Whittle P, Hogan T, Jenkins WD, Rietmeijer CA, Gaydos CA. Internet-based screening for sexually transmitted infections to reach nonclinic populations in the community: risk factors for infection in men. Sex Transm Dis. 2010 Dec;37(12):756-63. doi: 10.1097/OLQ.0b013e3181e3d771. PMID 20644498
- [Background] Gaydos CA, Barnes M, Aumakhan B, Quinn N, Agreda P, Whittle P, Hogan T. Can e-technology through the Internet be used as a new tool to address the Chlamydia trachomatis epidemic by home sampling and vaginal swabs? Sex Transm Dis. 2009 Sep;36(9):577-80. doi: 10.1097/OLQ.0b013e3181a7482f. No abstract available. PMID 19543145
- [Background] Gaydos CA, Dwyer K, Barnes M, Rizzo-Price PA, Wood BJ, Flemming T, Hogan MT. Internet-based screening for Chlamydia trachomatis to reach non-clinic populations with mailed self-administered vaginal swabs. Sex Transm Dis. 2006 Jul;33(7):451-7. doi: 10.1097/01.olq.0000200497.14326.fb. PMID 16652069
- [Derived] Patel AV, Abrams SM, Gaydos CA, Jett-Goheen M, Latkin CA, Rothman RE, Hsieh YH. Increasing HIV testing engagement through provision of home HIV self-testing kits for patients who decline testing in the emergency department: a pilot randomisation study. Sex Transm Infect. 2019 Aug;95(5):358-360. doi: 10.1136/sextrans-2018-053592. Epub 2018 Jun 14. PMID 29903889

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Self Testing Kit: This group will be provided a free Food and Drug Administration-approved HIV self-testing home kit (OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test). Participants in this group will also be provided 5 referral cards to give to their partners and peers in the drug, sex, and social networks for them to request a free HIV self-testing kit from the "I Want The Kit" website.
- No Intervention: No Self Testing Kit: This group will not receive a free Food and Drug Administration-approved HIV self-testing home kit (OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test). Participants in this group will not receive referral cards for their partners or peers for them to request a free HIV self-testing kit from the "I Want The Kit" website.
Period: Overall Study
Arm/Group | Experimental: Self Testing Kit | No Intervention: No Self Testing Kit
Started | 102 | 98
Completed | 63 | 72
Not Completed | 39 | 26
Not completed — Lost to Follow-up | 39 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Self Testing Kit | No Intervention: No Self Testing Kit | Total
Number analyzed (Participants) | 102 | 98 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 97 | 195
  >=65 years | 4 | 1 | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [24 to 42] | 38 [28 to 48] | 35 [25 to 45.5]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 39 | 37 | 76
  Female | 62 | 61 | 123
  Transgender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 81 | 85 | 166
  Unknown or Not Reported | 15 | 12 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 66 | 126
  White | 31 | 22 | 53
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 98 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Did HIV Testing
Description: Number of participants who did the HIV testing (HIV testing rate) will be determined by a telephone follow-up at 1 month after the index emergency department visit (enrollment).
Time Frame: At 1 month post enrollment
Population: 39 participants in Self Testing Kit group and 26 participants in No Self Testing Kit group were lost to follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Self Testing Kit: This group will be provided a free Food and Drug Administration-approved HIV self-testing home kit (OraQuick ADVANCE® Rapid HIV-1/2 Antibody Test). Participants in this group will also be provided 5 referral cards to give to their partners and peers in the drug, sex, and social networks for them to request a free HIV self-testing kit from the "I Want The Kit" website.
  HIV Self-testing
Arm/Group | Self Testing Kit | No Self Testing Kit
Number analyzed (Participants) | 63 | 72
Participants | 36 | 9

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Experimental: Self Testing Kit | No Intervention: No Self Testing Kit
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/98
Other Adverse Events (participants affected / at risk) | 0/102 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT03021005/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT03021005/ICF_001.pdf